CLINICAL TRIAL: NCT01996852
Title: Improving Erectile Function and Quality of Life After Prostate Cancer Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Premature terminated at institution request
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: The Cleveland Clinic (Other); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE14812; 05-12-05C (Other: University Hospitals at Case Medical Center Cancer IRB)
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer; Erectile Dysfunction Following Radical Prostatectomy; Erectile Dysfunction Following Simple Prostatectomy; Erectile Dysfunction
Keywords: Erectile dysfunction; ED; Prostate; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Standard ED Care (Active Comparator): Standard medical treatment of erectile dysfunction (ED) including administration of sildenafil citrate (Viagra) and/or vacuum constriction devices (pump)
  Interventions: Drug: sildenafil citrate; Device: Vacuum Constriction Device
- Standard ED Care + Cognitive-Behavioral Intervention (Experimental): standard medical treatment of ED (administration of sildenafil citrate (Viagra) and/or vacuum constriction devices (pump)) in addition to cognitive-behavioral meetings
  Interventions: Behavioral: Cognitive-behavioral Meetings; Drug: sildenafil citrate; Device: Vacuum Constriction Device
- Usual Care (UC) (No Intervention): Study participants will not receive any study intervention, but will continue with standard care.

INTERVENTIONS:
Behavioral: Cognitive-behavioral Meetings — The cognitive-behavioral intervention will consist of six monthly in-person meetings and five telephone follow-ups. In-person meetings include a 90-minute educational group session and five 60-minute therapeutic couple-based meetings which partners are asked to attend. The telephone follow-ups last 15-30 minutes and take place two weeks after each in-person meeting. They will review progress and provide support.
  Each monthly meeting has a focused topic: Introduction, Guided imagery, Sensate focus, Communication and relationship issues, and Review.
  Homework will be assigned at the end of each meeting. Generally, participants are instructed (a) practice guided imagery daily, (b) engage in sexual activity 1-2 times/ week after sildenafil intake and (c) use the pump every day for 10min.
  Arms: Standard ED Care + Cognitive-Behavioral Intervention
Drug: sildenafil citrate — 100mg of sildenafil citrate will be given twice a week to interested patients. Participants may start Sildenafil at a lower dose when needed.
  To increase external validity, participants will be given the choice of using Sildenafil in the study.
  Other Names: Viagra
  Arms: Standard ED Care; Standard ED Care + Cognitive-Behavioral Intervention
Device: Vacuum Constriction Device — The medical treatment entails a 10-minute daily use of VCD (pump).
  The VCD (pump) is a FDA approved marketing product and has a brochure and DVD that explain its usage. The clinical trials unit (CTU) nurse will dispense the VCD at the drug pick-up time and document it on a Device Accountability Form. The study coordinator has received manufacturer's training and can address questions that a subject may have about VCD on site or through a phone call.
  Other Names: VCD; Pump
  Arms: Standard ED Care; Standard ED Care + Cognitive-Behavioral Intervention

SUMMARY:
This is a research study of erectile dysfunction (ED) in men diagnosed with prostate cancer. 144 patients and partners will participate in the study. The purpose of this study is to test a new treatment that combines a cognitive-behavioral intervention with medication and a vacuum constrictive device to treat ED. This new treatment consists of multiple therapeutic elements that enhance compliance with medical treatment and increase sexual activity through enhancement of the sensual pleasure of sex and partner support.

DETAILED DESCRIPTION:
Erectile dysfunction (ED) is a common side effect of prostate cancer treatment. Existing medical treatment focuses on early penile rehabilitation, aiming to prevent penile shrinkage and preserve nerves and smooth muscles to facilitate erection return. It typically includes administration of phosphodiesterase type 5 inhibitor (PDE-5), application of vacuum constriction devices (VCD) or intracavernous injection immediately after prostate cancer treatment.

To evaluate the proposed intervention, a randomized, controlled longitudinal clinical trial will be conducted to examine the effect of this cognitive-behavioral intervention on early-stage prostate cancer patients with ED and their partners. The proposed study includes a pilot study, a randomized clinical trial (the main study) and data analysis. The study duration for main study participants is 10 months including one month of recruitment and baseline assessment, six months of intervention, and three months of follow-up. The study duration for pilot study participants is 7 months including one month of recruitment and baseline assessment plus six months of intervention.

The Pilot Study A pilot study will be conducted to develop and test the proposed study intervention over 12 months. The pilot study will recruit 36 early-stage prostate cancer patients and their partners. The 36 couples will be randomly assigned to three study arms: (1) standard medical treatment of ED (MED); (2) standard medical treatment of ED plus cognitive-behavioral intervention (MED+CBI); and (3) usual care (UC) in which the study participants will not receive any study intervention, but will continue with standard care that allows patient's request for ED treatment. The purpose to include the usual care group is to collect preliminary data to aid the estimation of intervention effect size, statistic power and sample size, and to compare the intervention outcome with the real world scenario in order to provide the justification for the inclusion or exclusion of the usual care arm in the main study. The pilot study participants will be assessed twice at baseline (T1) and 7 months (T2) only. Doppler Ultrasound of the penis will be performed at T1 and T2 to examine changes in the volume of penile blood flow in patients. Subjects are allowed to opt out of the Doppler Ultrasound test, because this pilot data is exploratory and five or more ultrasound tests per group are sufficient. Collecting and analyzing blood samples will be performed at T1 and T2 and subjects are allowed to opt out of this test as well. The blood sample will be collected in order to test transforming growth factor beta-1 (TGF-ß1) and to assess its relation to erectile function. The result will allow us to evaluate the intervention impact at molecular level and formulate a best possible intervention to ED.

The Main Study During a 4-year clinical trial study, 144 early-stage prostate cancer patients along with their partners will be randomly assigned to two study arms: (1) standard medical treatment of ED (MED) and (2) standard medical treatment of ED plus cognitive-behavioral intervention (MED+CBI). The MED includes administration of sildenafil citrate (Viagra) and/or vacuum constriction devices (pump). The MED+CBI entails six in-person sessions and five telephone follow-ups over six months. The patients will be assessed on erectile function (EF), quality of life (QOL) and mood at baseline (T1), 7 months (T2) and 10 months (T3). The partners will be assessed on QOL and mood at T1, T2 and T3. Doppler Ultrasound of the penis will be performed at T1 and T2 to examine changes in the volume of penile blood flow among 50 patients who will be consecutively selected from the two study groups, with 25 per study arm.

The long-term primary goals of the study are to:

1. Assess the effect of the new treatment on erection function, quality of life, and mood.
2. Assess the treatment compliance and frequency of sexual activity of the new treatment.
3. Investigate the mechanism in which the new treatment works.

The long-term secondary goals of the study are to:

1. Assess the effect of the new treatment on the quality of life and mood of the patient's partner.
2. Assess the changes in the volume of penile blood flow due to study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Stage I, II, and III prostate cancer
* Having completed definite treatment of localized prostate cancer (surgery or radiation);
* Presence of erectile dysfunction symptoms;
* Have a stable partner for six months who is willing to participate;
* Sexually active prior to cancer treatment (≥17 on the Sexual Health Inventory For Men- ("SHIM")).
* Prostatectomy with or without radiation for the pilot study patients only.

Exclusion Criteria:

* Receiving hormonal treatment;
* Cognitive impairment (≥5 on the Short Portable Mental Status Questionnaire (SPMSQ));
* Severe marital maladjustment that prevents a patient from benefiting from the proposed intervention (<85 on the Locke-Wallace Marital Adjustment Test);
* Taking nitrates of any kind;
* Congenital bleeding disorder or predisposition to priapism that is contraindicative to VCD use;
* Having untreated clinical depression and other psychotic mental disorders (e.g., bipolar, schizophrenia) (≥27 on the Center for Epidemiological Studies Depression Scale (CES-D)).
* Patients taking any potent inhibitor of cytochrome P450 3A4 (e.g., ketoconazole, itraconazole, erythromycin, etc).
* Patients taking concomitant alpha-adrenergic blocking agents.
* Patients with a clinically significant abnormality on screening ECG (taken within 12 weeks) that in the opinion of the investigator/co-investigator may increase the patient's cardiovascular risk in this study.
* Patients with a history of left ventricular outflow obstruction (e.g., aortic stenosis, idiopathic hypertrophic subaortic stenosis).
* Patients with a history of severely impaired autonomic control of blood pressure.
* Patients with resting hypotension (BP < 90/50 mm Hg), or resting hypertension (BP > 170/110 mm Hg) at Screening.
* Patients with known hypersensitivity to Sildenafil or other ingredients of Sildenafil.
* Patients with retinitis pigmentosa.
* Patients with active peptic ulceration.
* Patients who have previously experienced non-arteritic ischemic optic neuropathy (NAION).
* Patients taking other phosphodiesterase Type 5 (PDE5) inhibitors.
* Patients taking Coumadin, Pradaxa or other blood thinner drugs.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Zhang, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard ED Care: Standard medical treatment of erectile dysfunction (ED) including administration of sildenafil citrate (Viagra) and/or vacuum constriction devices (pump)
  sildenafil citrate: 100mg of sildenafil citrate will be given twice a week to interested patients. Participants may start Sildenafil at a lower dose when needed.
  To increase external validity, participants will be given the choice of using Sildenafil in the study.
  Vacuum Constriction Device: The medical treatment entails a 10-minute daily use of VCD (pump).
  The VCD (pump) is a FDA approved marketing product and has a brochure and DVD that explain its usage. The clinical trials unit (CTU) nurse will dispense the VCD at the drug pick-up time and document it on a Device Accountability Form. The study coordinator has received manufacturer's training and can address questions that a subject may have about VCD on site or through a phone call.
- Standard ED Care + Cognitive-Behavioral Intervention: standard medical treatment of ED (administration of sildenafil citrate (Viagra) and/or vacuum constriction devices (pump)) in addition to cognitive-behavioral meetings
  Cognitive-behavioral Meetings: The cognitive-behavioral intervention will consist of six monthly in-person meetings and five telephone follow-ups. In-person meetings include a 90-minute educational group session and five 60-minute therapeutic couple-based meetings which partners are asked to attend. The telephone follow-ups last 15-30 minutes and take place two weeks after each in-person meeting. They will review progress and provide support.
  Each monthly meeting has a focused topic: Introduction, Guided imagery, Sensate focus, Communication and relationship issues, and Review.
  Homework will be assigned at the end of each meeting. Generally, participants are instructed (a) practice guided imagery daily, (b) engage in sexual activity 1-2 times/ week after sildenafil intake and (c) use the pump every day for 10min.
Period: Overall Study
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated prematurely by the IRB. As per the IRB determination, data are not accessible to the study team for reporting.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC) | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Erectile Function Improvement
Description: Change in Total score in the International Index of Erectile Function (IIEF) between baseline and 10 months. The IIEF assesses male sexual function in five domains: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. Higher scores indicate improved functioning.
Time Frame: 10 months after start of treatment
Population: as for baseline characteristics
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Change in Number of Erections
Description: Change from baseline in the number of patients with a score of >=22 on the International Index of Erectile Function (IIEF). This score signifies the presence of erection.
Time Frame: 10 months after start of treatment
Population: as for baseline characteristics
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Erectile Function Improvement
Description: Change in Total score in the International Index of Erectile Function (IIEF) between baseline and 7 months. The IIEF assesses male sexual function in five domains: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. Higher scores indicate improved functioning.
Time Frame: 7 months after start of treatment
Population: as for baseline characteristics
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Change in Number of Erections
Description: as for outcome 2
Time Frame: 7 months after start of treatment
Population: as for baseline characteristics
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Sexual Quality of Life (QoL) Improvement
Description: Change from baseline in the total score of the Sexual Quality of Life (male/female) scales. Higher scores indicate better quality of life.
Time Frame: 10 months after start of treatment
Population: as for baseline characteristics
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in Overall Quality of Life (QoL) Score
Description: Change in the total score from baseline on the Short-Form-36 Health Survey (SF36) will be used to show changes in QoL. Higher scores indicate increased QoL. QOL in eight dimensions, including physical, role and social functioning, role limitations, and general physical and mental health.
Time Frame: 10 months after start of treatment
Population: as for baseline characteristics
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Improved Mood Score
Description: Change from baseline in the sub-score from the 21-item Profile of Mood States (POMS) will be used to measure psychological adjustment to cancer. It will be used to measure depression, anxiety and anger. Higher scores indicate more mood disorder.
Time Frame: 10 months after start of treatment
Population: as for baseline characteristics
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change in Treatment Compliance
Description: Change from baseline in the number of patients compliant with treatment. Patients will be described as regular user, intermittent user, or drop out based on the information recorded in the patients Sex Diary over the previous seven days.
Time Frame: 10 months after start of treatment
Population: as for baseline characteristics
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change in Frequency of Sexual Activity
Description: Change from baseline in the mean value of sexual activities ((1) Sexual encounters; (2) Sexual simulation; (3) intercourse; and (ejaculation)) experienced by each participant over the previous seven days
Time Frame: 7 months after start of treatment
Population: as for baseline characteristics
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Change in Frequency of Sexual Activity
Description: as for outcome 9
Time Frame: 10 months after start of treatment
Population: as for baseline characteristics
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change in Treatment Compliance
Description: as for outcome 8
Time Frame: 7 months after start of treatment
Population: as for baseline characteristics
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Sexual Quality of Life (QoL) Improvement
Description: Change from baseline in the total score of the Sexual Quality of Life (male/female) scales
Time Frame: 7 months after start of treatment
Population: as for baseline characteristics
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Change in Overall Quality of Life (QoL) Score
Description: as for outcome 6
Time Frame: 7 months after start of treatment
Population: as for baseline characteristics
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
Number analyzed (Participants) | 0 | 0 | 0

14. Other Pre Specified Outcome: Self-Efficacy Improvement
Description: Change from baseline in the mean score of Bandura's measure to assess self-efficacy. This scale is scored from 0-100, where 100 indicates complete confidence.
Time Frame: 7 months after start of treatment
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Self-Efficacy Improvement
Description: as for outcome 14
Time Frame: 10 months after start of treatment
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in Level of Sensual Pleasure of Sex
Description: Change from baseline in a sub-score of the Sexual Function Questionnaire where higher scores indicate greater pleasure.
Time Frame: 7 months after start of treatment
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in Level of Sensual Pleasure of Sex
Description: Change from baseline in a sub-score of the Sexual Function Questionnaire where higher scores indicate greater pleasure.
Time Frame: 10 months after start of treatment
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Change in Perceived Partner Support
Description: change from baseline in a total score from a sub-scale of the Social Support for Exercise Behavior Questionnaire as modified by the study team to measure partner support for rehabilitation. Higher scores will indicate greater support.
Time Frame: 7 months after start of treatment
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change in Perceived Partner Support
Description: as for outcome 18
Time Frame: 10 months after start of treatment
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Change in Flaccid Penile Length
Description: Change from baseline in the total length of patients flaccid penis. Length will be measured using Mounding's method
Time Frame: 7 months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Change in Flaccid Penile Length
Description: Change from baseline in the total length of patients flaccid penis. Length will be measured using Mounding's method
Time Frame: 10 months
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Change in Stretched Penile Length
Description: Change from baseline in the total length of patients stretched penis. Length will be measured using Mounding's method
Time Frame: 7 months
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Change in Stretched Penile Length
Description: Change from baseline in the total length of patients stretched penis. Length will be measured using Mounding's method
Time Frame: 10 months
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Change in Volume of Flaccid Penile Blood Flow
Description: Change from baseline in the total penile blood flow will be assessed by a color and spectral Doppler ultra sound of the cavernosal arteries
Time Frame: 7 months after start of treatment
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Change in Volume of Flaccid Penile Blood Flow
Description: as for outcome 24
Time Frame: 10 months after start of treatment
Reporting Status: Not Posted

26. Other Pre Specified Outcome: TGF-B1 Levels
Description: Total level of Transforming Growth Factor Beta-1 levels will be assessed using a commercially available assay
Time Frame: baseline - 1 week after start of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The study was terminated prematurely by the IRB. As per the IRB determination, data are not accessible to the study team for reporting.
Description: The study was terminated prematurely by the IRB. As per the IRB determination, data are not accessible to the study team for reporting.
Arm/Group | Standard ED Care | Standard ED Care + Cognitive-Behavioral Intervention | Usual Care (UC)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely by the IRB. As per the IRB determination, data are not accessible to the study team for reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes